CLINICAL TRIAL: NCT01250587
Title: A Dose-Escalating Phase I Study to Evaluate the Safety, Pharmacokinetics and Efficacy of PDC31 in Patients With Primary Dysmenorrhea
Brief Title: Dose-Finding Study of PDC31 in Patients With Primary Dysmenorrhea
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PDC Biotech GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PDC-3111
Record Dates: First submitted 2010-11-29; First posted 2010-12-01 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-09

CONDITIONS: Dysmenorrhea
Keywords: Open label; dose-finding Phase 1 study
MeSH Terms: conditions — Dysmenorrhea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PDC31 (Experimental)
  Interventions: Drug: PDC31

INTERVENTIONS:
Drug: PDC31 — This study involves the sequential administration of PDC31 to 4 cohorts of patients. The dose will be escalated in the absence of dose-limiting toxicities. PDC31 is to be administered as a 3-hour continuous infusion.

SUMMARY:
The purpose of this study is to determine a safe and effective dose range for intravenous administration (infusion) of PDC31 by determining the maximum tolerated dose of PDC31 in patients with primary dysmenorrhea.

DETAILED DESCRIPTION:
This is an open-label, multi-centre, dose-escalating first-in-human Phase I study of PDC31 in patients with primary dysmenorrhea aimed at determining the maximum tolerated dose (MTD) of PDC31 in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Otherwise healthy females with a history of primary dysmenorrhea
* Using effective birth control excluding intrauterine contraceptive device (IUCD)
* Must be 18 years of age or older
* Must give written informed consent to participate in this study

Exclusion Criteria:

* Patients with an intrauterine contraceptive device or using oral contraceptives within 3 months of treatment in this study
* Patients with confirmed pelvic inflammatory disease, endometriosis or adenomyosis
* Patients who are pregnant or who test positive at baseline or are at risk of becoming pregnant while on study
* Patients who are breastfeeding
* Patients with hepatic or renal function tests greater than the upper limit of normal and deemed clinically significant by the Investigator at screening
* Patients with a clinically significant medical or psychiatric disorder or a serious medical conditions within the past 6 months which in the opinion of the investigator, should prohibit participation in this study
* Patients who have been exposure to any investigational drug within 4 weeks prior to screening

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-11; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Occurrence of Dose-Limiting Toxicity | Observed following PDC31 administration to 30 day follow-up

SECONDARY OUTCOMES:
Pharmacokinetic profiling of PDC31 and pharmacodynamic effects of PDC31 as observed on uterine contractility | Observed immediately following PDC31 administration

CONTACTS AND LOCATIONS:
Locations (4):
- Austria (2):
  - Innsbruck Medical University, Innsbruck
  - Medical University of Vienna, Vienna
- Germany (2):
  - University Hospital Hamburg-Eppendorf, Hamburg
  - University of Mainz, Mainz

REFERENCES:
- [Derived] Bottcher B, Laterza RM, Wildt L, Seufert RJ, Buhling KJ, Singer CF, Hill W, Griffin P, Jilma B, Schulz M, Smith RP. A first-in-human study of PDC31 (prostaglandin F2alpha receptor inhibitor) in primary dysmenorrhea. Hum Reprod. 2014 Nov;29(11):2465-73. doi: 10.1093/humrep/deu205. Epub 2014 Aug 27. PMID 25164021